CLINICAL TRIAL: NCT00471185
Title: Oral Administration of the GnRH Antagonist Acyline in Normal Men
Brief Title: ACY-6 Oral Administration of Acyline
Acronym: ACY-6
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Merrion Pharmaceuticals, LLC (Industry)
Responsible Party: John K Amory, MD, MPH, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31511-W; 07-4947-W 02 (Other: UW Human Subjects Division)
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Contraception
Keywords: Male Contraception; Acyline
MeSH Terms: interventions — acyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Subjects will receive progressively increasing doses of 10, 20 and 40 mg of oral acyline, on 3 occasions, each separated by 1 week
  Interventions: Drug: Acyline

INTERVENTIONS:
Drug: Acyline — 10, 20 and 40 mg of Oral acyline, given on 3 occasions, separated by 1 week.

SUMMARY:
In this study, we propose oral dosing of GIPET enhanced oral acyline (MER-104) to determine if this potentially useful compound is safe and effective at suppression of gonadotropins after oral dosing in man.

Hypothesis: A single dose of Acyline will suppress gonadotropins, and testosterone, estradiol and dihydrotestosterone (DHT) for 24 hours in man, and the magnitude and duration of the suppression will increase with increasing doses of Acyline.

DETAILED DESCRIPTION:
The purpose of this study is to test how the body responds to a new oral form of acyline and to also look at the safety of oral acyline.

Acyline temporarily blocks the production of the hormone testosterone in normal men. It has been given to over 100 men in an injection form. This study will be testing acyline in a pill form. This is the first time the pill form has been tested in humans.

This study may help develop an oral form of a testosterone-blocker, which may be useful in the treatment of diseases such as prostate cancer, premature puberty and possibly in a male contraceptive.

This study requires three 12-hour blood draw periods for pharmacokinetics (PK) testing. PK testing looks to see how much study drug is in the blood. This gives information about how the body handles and gets rid of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18-50 years of Age in good health

Exclusion Criteria:

* Men in poor health, significant chronic or acute medical illness, known history of alcohol, illicit drug or anabolic steroid abuse

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the suppressive effects of GIPET-enhanced oral Acyline on pituitary gonadotropin and testosterone secretion in normal men and to assess any potential side effects of GIPET enhanced oral Acyline | 28-days

SECONDARY OUTCOMES:
To define the pharmacokinetics of GIPET enhanced oral Acyline | 28-days
Assess any potential side effects of GIPET enhanced oral Acyline | 28-days

CONTACTS AND LOCATIONS:
Overall Officials: John K Amory, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Herbst KL, Anawalt BD, Amory JK, Bremner WJ. Acyline: the first study in humans of a potent, new gonadotropin-releasing hormone antagonist. J Clin Endocrinol Metab. 2002 Jul;87(7):3215-20. doi: 10.1210/jcem.87.7.8675. PMID 12107227
- [Background] Herbst KL, Coviello AD, Page S, Amory JK, Anawalt BD, Bremner WJ. A single dose of the potent gonadotropin-releasing hormone antagonist acyline suppresses gonadotropins and testosterone for 2 weeks in healthy young men. J Clin Endocrinol Metab. 2004 Dec;89(12):5959-65. doi: 10.1210/jc.2003-032123. PMID 15579744
- [Background] Matthiesson KL, Amory JK, Berger R, Ugoni A, McLachlan RI, Bremner WJ. Novel male hormonal contraceptive combinations: the hormonal and spermatogenic effects of testosterone and levonorgestrel combined with a 5alpha-reductase inhibitor or gonadotropin-releasing hormone antagonist. J Clin Endocrinol Metab. 2005 Jan;90(1):91-7. doi: 10.1210/jc.2004-1228. Epub 2004 Oct 27. PMID 15509637
- [Background] Amory JK, Bremner WJ. Oral testosterone in oil plus dutasteride in men: a pharmacokinetic study. J Clin Endocrinol Metab. 2005 May;90(5):2610-7. doi: 10.1210/jc.2004-1221. Epub 2005 Feb 15. PMID 15713724
- [Background] Amory JK, Page ST, Bremner WJ. Oral testosterone in oil: pharmacokinetic effects of 5alpha reduction by finasteride or dutasteride and food intake in men. J Androl. 2006 Jan-Feb;27(1):72-8. doi: 10.2164/jandrol.05058. PMID 16400081
- [Background] Page ST, Lin DW, Mostaghel EA, Hess DL, True LD, Amory JK, Nelson PS, Matsumoto AM, Bremner WJ. Persistent intraprostatic androgen concentrations after medical castration in healthy men. J Clin Endocrinol Metab. 2006 Oct;91(10):3850-6. doi: 10.1210/jc.2006-0968. Epub 2006 Aug 1. PMID 16882745
- [Background] Page ST, Amory JK, Anawalt BD, Irwig MS, Brockenbrough AT, Matsumoto AM, Bremner WJ. Testosterone gel combined with depomedroxyprogesterone acetate is an effective male hormonal contraceptive regimen and is not enhanced by the addition of a GnRH antagonist. J Clin Endocrinol Metab. 2006 Nov;91(11):4374-80. doi: 10.1210/jc.2006-1411. Epub 2006 Aug 29. PMID 16940442
- [Result] Snyder CN, Clark RV, Caricofe RB, Bush MA, Roth MY, Page ST, Bremner WJ, Amory JK. Pharmacokinetics of 2 novel formulations of modified-release oral testosterone alone and with finasteride in normal men with experimental hypogonadism. J Androl. 2010 Nov-Dec;31(6):527-35. doi: 10.2164/jandrol.109.009746. Epub 2010 Apr 8. PMID 20378927